CLINICAL TRIAL: NCT04577872
Title: The Effect of Pelvic Floor Exercise on Urinary Incontinence and Quality of Sex Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 019234/2014/OTIG
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-09

CONDITIONS: Pelvic Floor Muscle Weakness; Urinary Incontinence
Keywords: pelvic floor muscle training; transverse abdominal muscle; ultrasound measurement; urinary incontinence; vaginal surface electromyography
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine group (n=22) (Experimental): The 22 participants with lower muscle strength (under 60 microvolt) comprised the supine group.
  Interventions: Other: Pelvic floor muscle training
- Sitting group (n=19) (Experimental): The 19 participants with higher muscle strength (over 60 microvolt) formed the sitting group.
  Interventions: Other: Pelvic floor muscle training
- Control group (n=14) (No Intervention): The control group comprised 7 individuals with lower muscle strength (under 60 microvolt) and 7 with higher muscle strength (over 60 microvolt)

INTERVENTIONS:
Other: Pelvic floor muscle training — The treatment for the sitting group comprised 8 sessions, with a 1-hour combined pelvic floor muscle training (cPFM-T) session each week in a group and 15 minutes of individual home training, six times a week for a total of 8 weeks of treatment. All training sessions comprised warming-up, gradual muscle strengthening and relaxation exercises. In the study, before and after the training programme, we used a self-administered questionnaire.We measured changes in pelvic floor muscle activity with a vaginal surface electromyographic instrument. We performed the transversus abdominis measurements at the same time as the vaginal measurements and pelvic floor muscle tasks.
  Arms: Sitting group (n=19); Supine group (n=22)

SUMMARY:
This physiotherapist-guided group training programme should be performed in both the supine and the sitting positions; it is investigated, which is better and more cost-effective in patient motivation.

DETAILED DESCRIPTION:
Here we aimed to investigate whether-based on trunk muscle synergism-the condition and functioning of the pelvic floor muscle would improve in the sitting and supine postures or in the control group during pelvic floor muscle training with forced exhalation. We enrolled nulliparous women in supine (n = 22), sitting (n = 19) and control (n = 14) groups. We performed the 8-week combined pelvic floor muscle training programme. We examined the effect of training on the parameters with the Kruskal-Wallis test, and the pairwise comparisons with the Mann-Whitney U-test and the Wilcoxon-rank test with the Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* We included in the study groups women participants willing to participate in the study and able to contract the pelvic floor and transversus abdominis muscles correctly. Participants were required to maintain their everyday activities (attending lessons, sport activities, and so on).

Exclusion Criteria:

* known neurological or rheumatological diseases and previous vaginal or abdominal surgery.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — nulliparous women
Enrollment: 55 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Investigation of the effects of the pelvic floor muscle training (PFM-T) | 28 months
  It is measured the change of the pelvic floor muscle with Vaginal surface electromyography (vsEMG).

CONTACTS AND LOCATIONS:
Overall Officials: Edit Nagy, Habil. PhD, Principal Investigator — University of Szeged, Faculty of Health Sciences and Social Studies

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madill SJ, McLean L. Quantification of abdominal and pelvic floor muscle synergies in response to voluntary pelvic floor muscle contractions. J Electromyogr Kinesiol. 2008 Dec;18(6):955-64. doi: 10.1016/j.jelekin.2007.05.001. Epub 2007 Jul 23. PMID 17646112
- [Background] Chmielewska D, Stania M, Sobota G, Kwasna K, Blaszczak E, Taradaj J, Juras G. Impact of different body positions on bioelectrical activity of the pelvic floor muscles in nulliparous continent women. Biomed Res Int. 2015;2015:905897. doi: 10.1155/2015/905897. Epub 2015 Feb 22. PMID 25793212
- [Result] Haslam J. The prevalence of stress urinary incontinence in women. Nurs Times. 2004 May 18;100(20):71-3. No abstract available. PMID 15176284
- [Result] KEGEL AH. Progressive resistance exercise in the functional restoration of the perineal muscles. Am J Obstet Gynecol. 1948 Aug;56(2):238-48. doi: 10.1016/0002-9378(48)90266-x. No abstract available. PMID 18877152
- [Result] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Result] Capson AC, Nashed J, Mclean L. The role of lumbopelvic posture in pelvic floor muscle activation in continent women. J Electromyogr Kinesiol. 2011 Feb;21(1):166-77. doi: 10.1016/j.jelekin.2010.07.017. Epub 2010 Sep 15. PMID 20833070
- [Result] Sapsford RR, Richardson CA, Stanton WR. Sitting posture affects pelvic floor muscle activity in parous women: an observational study. Aust J Physiother. 2006;52(3):219-22. doi: 10.1016/s0004-9514(06)70031-9. PMID 16942457
- See also: Related Info — http://www.medrxiv.org/content/10.1101/2020.03.20.20039586v1

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-04-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04577872/Prot_SAP_ICF_000.pdf